CLINICAL TRIAL: NCT01409330
Title: Short Term Diet Intervention in Newly Diagnosed Type 2 Diabetes. a Randomised, Multicentric, Controlled, Clinical Trial
Brief Title: German Diabetes-Diet-Intervention and Energy Restriction-Trial (DDIET)
Acronym: DDIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DDIET3521
Record Dates: First submitted 2011-06-08; First posted 2011-08-04 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: insulin sensitivity; type 2 diabetes; diet intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypocaloric diet containing increased fibers and coffee (Experimental): In the intervention group the patients are allowed to eat only white meat and fish. They also need to increase their daily fiber intake to 50grams and drink 5 cups of coffee a day.
  Interventions: Dietary Supplement: diet intervention
- hypocaloric diet containing red meat (Active Comparator): control group (n=20): diet according to the ADA/EASD guidelines (50% carbohydrates, 20% proteins, 30% fat). In the control group the patients should eat 150 grams of red meat a day and are not allowed to consume alcohol, coffee and whole grains.
  Interventions: Dietary Supplement: diet intervention

INTERVENTIONS:
Dietary Supplement: diet intervention — 8-week diet lacking red meat, but containing increased fibers and coffee (verum) versus standard recommendation (control) eating red meat.

SUMMARY:
Diet intervention according to the German Diabetes Risk Score in newly diagnosed type 2 diabetes.

This study aims to explore the effect of diet lacking red meat, but containing increased fibers and coffee (verum) versus standard recommendation (control) in a multicenter setting.

DETAILED DESCRIPTION:
This study is a randomised, multicenter controlled trial Our Aim is to test the effects of an 8-week diet lacking red meat, containing increased fibers and coffee (verum) versus standard recommendation (control)in a multicenter setting.

We are expecting that the verum diet will improve insulin sensitivity and insulin secretion due to reductions in visceral and hepatic fat along with improved adipocyte cytokine secretion profiles

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* disease duration for five years or less,
* age of 69 years or less,
* body mass index of 30 kg/m2 or more,
* hemoglobin A1c of 5,5 % to 9%
* patient should be on standard diet or metformin +/- acarbose monotherapy
* patient should be without exclusion criteria for coffee consumption

Exclusion Criteria:

* disease duration more than five years,
* age of > 69 years,
* body mass index of < 30 kg/m2,
* hemoglobin A1c < 5,5 % or > 9%
* if patient becomes insulin therapy
* if patient has exclusion criteria for coffee consumption
* if patient is non-compliant with study protocol
* if patient is pregnant
* if patient has acute infection
* if patient has anaemia
* if patient has malignancies
* if patient has autoimmune or immune compromising diseases including HIV/AIDS
* if patient has psychiatric diseases or addiction

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
whole body insulin sensitivity | 8 weeks
  measurement of whole body insulin sensitivity with hyperinsulinamic euglicamic clamp

SECONDARY OUTCOMES:
total body fat | 8 weeks
  MRI measurement of the effects of 8-week diet intervention on total body fat
intramyocellular lipids | 8 weeks
  MRS measurement to investigate the effects of diet intervention on ectopic lipid content in skeletal muscle
skeletal muscle mitochondrial function - insulin signaling | 8 weeks
  muscle biopsy for assessment of insulin signaling
hepatocellular lipids | 8 weeks
  MRS measurement to investigate the effects of diet intervention on ectopic lipid content in liver(HCL)
skeletal muscle mitochondrial function - phosphate-recovery time | 8 weeks
  skeletal muscle mitochondrial function in vivo assessed as phosphate-recovery time with MRS
insulin secretion | 8 weeks
  measurement of insulin secretion with glucagon test, mixed-meal test and intravenous glucose tolerance test
pancreatic fat | 8 weeks
  MRI measurement of the effects of 8-week diet intervention on pancreatic fat

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Study Director — German Diabetes Center
Locations (6):
- Germany (6):
  - German Diabetes Center, Düsseldorf, North Rhine-Westphalia
  - Charite, Department of Internal Medicine, Berlin
  - University Hospital, Department of Internal Medicine III, Dresden
  - University Hospital, Department of Internal Medicine I, Heidelberg
  - Klinikum der Universität München (KUM), Munich
  - University Hospital, Department of Internal Medicine IV, Tübingen

REFERENCES:
- [Derived] Pafili K, Zaharia OP, Strassburger K, Knebel B, Herder C, Huttasch M, Karusheva Y, Kabisch S, Strom A, Nowotny B, Szendroedi J, Roden M. PNPLA3 gene variation modulates diet-induced improvement in liver lipid content in type 2 diabetes. Clin Nutr. 2025 May;48:6-15. doi: 10.1016/j.clnu.2025.02.032. Epub 2025 Mar 6. PMID 40090039
- [Derived] Karusheva Y, Kunstein L, Bierwagen A, Nowotny B, Kabisch S, Groener JB, Fleitmann AK, Herder C, Pacini G, Strassburger K, Haring HU, Nawroth PP, Pfeiffer AFH, Burkart V, Mussig K, Roden M, Szendroedi J. An 8-week diet high in cereal fiber and coffee but free of red meat does not improve beta-cell function in patients with type 2 diabetes mellitus: a randomized controlled trial. Nutr Metab (Lond). 2018 Dec 29;15:90. doi: 10.1186/s12986-018-0324-5. eCollection 2018. PMID 30619502
- [Derived] Ziegler D, Strom A, Nowotny B, Zahiragic L, Nowotny PJ, Carstensen-Kirberg M, Herder C, Roden M. Effect of Low-Energy Diets Differing in Fiber, Red Meat, and Coffee Intake on Cardiac Autonomic Function in Obese Individuals With Type 2 Diabetes. Diabetes Care. 2015 Sep;38(9):1750-7. doi: 10.2337/dc15-0466. Epub 2015 Jun 12. PMID 26070589
- [Derived] Nowotny B, Zahiragic L, Bierwagen A, Kabisch S, Groener JB, Nowotny PJ, Fleitmann AK, Herder C, Pacini G, Erlund I, Landberg R, Haering HU, Pfeiffer AF, Nawroth PP, Roden M. Low-energy diets differing in fibre, red meat and coffee intake equally improve insulin sensitivity in type 2 diabetes: a randomised feasibility trial. Diabetologia. 2015 Feb;58(2):255-64. doi: 10.1007/s00125-014-3457-8. Epub 2014 Nov 26. PMID 25425219